CLINICAL TRIAL: NCT05949905
Title: Efficacy of a Stage-matched Intervention Based on Transtheoretical Model of Change in Changing the Digital Gaming Behavior Among Male High School Students: A Randomized Controlled Trial
Brief Title: A Stage-matched Intervention Based on Transtheoretical Model of Change in Changing the Videogaming Behavior
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Collaborators: Melak Obaid Nghaimesh (Unknown)
Responsible Party: Principal Investigator, Mohammed Baqer Habeeb Abd Ali, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: Digital Gaming Behavior
Record Dates: First submitted 2023-06-28; First posted 2023-07-18 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Video Game Addiction
Keywords: High school students; Problematic digital gaming; Transtheoretical Model of Change
MeSH Terms: conditions — Technology Addiction

STUDY DESIGN:
Who Masked: Participant
Masking Description: The researchers will use two groups (study and control) in which participants will be randomly selected and assigned in each of the study and control groups using simple random sampling.
  The study intervention will be designed based on each Stage of Change of the Transtheoretical Model of Change in that participants in each Stage of Change will receive the intervention that matches the Stage of Change they would be in.
  A 12-week interval would be considered between administering the intervention and posttest 1 and the same interval would be used between posttest 1 and posttest 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Precontemplation, Contemplation, Preparation, Action, and Maintenance-based intervention (Experimental): The intervention that would consider the Processes of Change that people use when they would be in the Precontemplation Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Contemplation-based intervention (Experimental): The intervention that would consider the Processes of Change that people use when they would be in the Contemplation Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Preparation-based intervention (Experimental): The intervention that would consider the Processes of Change that people use when they would be in the Preparation Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Action-based intervention (Experimental): The intervention that would consider the Processes of Change that people use when they would be in the Action Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Maintenance-based intervention (Experimental): The intervention that would consider the Processes of Change that people use when they would be in the Maintenance Stage of Change.
  Interventions: Behavioral: Stage-matched interventions

INTERVENTIONS:
Behavioral: Stage-matched interventions — The intervention would be using the Processes of Change that match each Stage of Change.

SUMMARY:
A Stage-matched randomized controlled trial seeks to change the problematic digital gaming behavior among high school male students.

DETAILED DESCRIPTION:
The researchers will use two groups (study and control) in which participants will be randomly selected and assigned in each of the study and control groups using simple random sampling.

The study intervention will be designed based on each Stage of Change of the Transtheoretical Model of Change in that participants in each Stage of Change will receive the intervention that matches the Stage of Change they would be in.

A 12-week interval would be considered between administering the intervention and posttest 1 and the same interval would be used between posttest 1 and posttest 2.

ELIGIBILITY:
Inclusion Criteria:

* High school male students who do not experience any psychiatric-mental disorder.

Exclusion Criteria:

* High school male students who experience any psychiatric-mental disorder.

Ages: 15 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — High school male students who do not experience any psychiatric-mental disorder.
Enrollment: 144 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Stages of Change Scale for Digital Gaming Behavior | 6 months
  Stages of Change Scale for Digital Gaming Behavior that measures individuals' readiness to avoid problematic digital gaming behavior

CONTACTS AND LOCATIONS:
Locations (1):
- University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided